CLINICAL TRIAL: NCT05786508
Title: Partners for Pain & Wellbeing Equity: A Randomized Trial of Community Supported Complementary and Integrative Health Self-management for Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R61AT012309 (NIH); 1R61AT012309 (NIH)
Record Dates: First submitted 2023-02-15; First posted 2023-03-27 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Neck Pain; Low Back Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partners4Pain program (Experimental): adults with chronic neck or back pain from populations that experience health disparities due to race/ethnicity or socioeconomic status
  Interventions: Other: Partners4Pain program
- Key to Wellbeing program (Active Comparator): adults with chronic neck or back pain from populations that experience health disparities due to race/ethnicity or socioeconomic status
  Interventions: Other: Key to Wellbeing program

INTERVENTIONS:
Other: Partners4Pain program — Partners4Pain is a self-management program of evidence based complementary and integrative health approaches for pain including pain education, mindfulness, cognitive behavioral approaches, and neck/back specific exercises.
  The intervention program will include nine, 90-minute group sessions that occur weekly for 9 weeks
  Arms: Partners4Pain program
Other: Key to Wellbeing program — Keys to Wellbeing is a general health and wellbeing education program addressing topics such as keeping socially connected, finding meaning and purpose, addressing mental health, and keeping physically fit. The program was designed to control for time, attention, and many other key contextual factors (e.g., program format, materials).
  The intervention program will include nine, 90-minute group sessions that occur weekly for 9 weeks
  Arms: Key to Wellbeing program

SUMMARY:
The focus of this project is on developing and optimizing community-based programs for the self-management of back or neck pain for individuals from populations that experience health disparities (BP-PEHD). Community-engaged research approach will be used to conduct quality improvement activities that involves gathering feedback from multiple stakeholders to inform development of the study interventions and materials which will be followed by a randomized pilot study to evaluate feasibility.

Supported by the National Center for Complementary and Integrative Health through the National Institutes of Health's HEAL initiative (https://heal.nih.gov/)"

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed and dated informed consent form
* State willingness to comply with all study procedures outlined in the consent form
* Be 18 years of age or older
* Have self-reported chronic back pain (defined as pain in the low or mid back, or neck pain) which has lasted for 3 months or longer
* Have a score of 3 or higher on the self-reported Pain, Enjoyment of Life and General Activity (PEG) scale (0 to 10)
* Be a member of one or more of the following NIH-designated health disparity populations: American Indian/Alaska Native, Asian, Black/African American, Hispanic/Latino, Native Hawaiian/Pacific Islanders, Socioeconomically disadvantaged (annual household income less than $50,000)

Exclusion Criteria:

* Hospitalization for severe mental illness in past six months because the mindfulness and behavioral mind-body practices (e.g., meditation, progressive muscle relaxation, etc.) in the experimental intervention may aggravate symptoms of severe mental illness
* Active psychotic symptoms, suicidal ideation, or manic episodes in the past three months for the same reasons noted in #1
* Self-reported cancer with active treatment involving radiation or chemotherapy due to the potential for complications of their back or neck pain and impact on health outcomes
* Dementia - Mini Mental State Exam score of 23 or lower for those with suspicion of cognitive impairment due to safety risks (e.g., not being able to follow directions for safe physical exercise)
* Self-reported pregnancy due to the fact that back pain is often associated with pregnancy and differs from non-pregnancy related back pain and thus might have different impacts on health outcomes
* Children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roni Evans, PhD, DC,MS, Principal Investigator — University of Minnesota; Brent Leininger, PhD, DC, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Partners4Pain Program: Partners4Pain is a self-management program of evidence based complementary and integrative health approaches for pain including pain education, mindfulness, cognitive behavioral approaches, and neck/back specific exercises. The intervention program included nine, 90-minute group sessions that occurred weekly for 9 weeks
- Key to Wellbeing Program: Keys to Wellbeing is a general health and wellbeing education program addressing topics such as keeping socially connected, finding meaning and purpose, addressing mental health, and keeping physically fit. The program was designed to control for time, attention, and many other key contextual factors (e.g., program format, materials). The intervention program included nine, 90-minute group sessions that occurred weekly for 9 weeks
Period: Overall Study
Arm/Group | Partners4Pain Program | Key to Wellbeing Program
Started | 26 | 25
Completed | 24 | 25
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Partners4Pain Program | Key to Wellbeing Program | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13.5) | 57 (15.9) | 56 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 6 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity using 2020 U.S. census questionnaire
  Participants
    No Hispanic, Latino, or Spanish origin | 23 | 22 | 45
    Mexican, Mexican American, Chicano | 1 | 1 | 2
    Another Hispanic, Latino, or Spanish origin (e.g. Savadorian, Dominican, Columbian, Guatemalan, etc) | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race using 2020 U.S. census questionnaire
  Participants
    Black or African American (African American, Jamaican, Haitian, Nigerian, Ethiopian, Somali, etc.) | 16 | 13 | 29
    White (German, Irish, English, Italian, Lebanese, Egyptian, etc.) | 5 | 7 | 12
    Chinese | 2 | 0 | 2
    Asian Indian | 1 | 0 | 1
    Other Asian (Pakistani, Cambodian, Hmong, etc.) | 0 | 1 | 1
    American Indian or Alaska Native | 0 | 1 | 1
    Other Race (Mestizo) | 0 | 1 | 1
    Other Race (Mexican) | 1 | 0 | 1
    More Than One Race | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51
Pain, Enjoyment of Life and General Activity (PEG) [Mean (Standard Deviation); unit: units on a scale] — Three questions about the past week's pain. One question asks about pain severity and two questions ask about pain interference. Each item is rated on a 0-10 scale. Responses are added together and divided by three to get a final score ranging from 0 to 10. A higher score indicates more severe pain and pain-related interference with life and activities.
  units on a scale | 6.7 (2.2) | 6.4 (1.7) | 6.5 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility: # of Enrolled Participants
Description: Demonstrate the ability to recruit and retain subjects in the clinical study as follows: Randomize at least 30 participants
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Participants: Individuals enrolled into the randomized trial
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 51
Participants | 51

2. Primary Outcome: Recruitment Feasibility: % of Enrolled Participants From NIH-defined Racial or Ethnic Disparity Groups
Description: Demonstrate the ability to recruit and retain subjects in the clinical study as follows: 75% or more of randomized participants are from NIH-defined racial/ethnic health disparity groups;
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 51
Participants | 40

3. Primary Outcome: Participant Retention Feasibility: Primary Outcome Measurement
Description: Demonstrate the ability to recruit and retain subjects in the clinical study as follows: 80% or more of randomized participants are retained for primary outcome measurement at the end of the study (2 month follow up) regardless of adherence to the intervention
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 51
Participants | 49

4. Primary Outcome: Intervention Delivery Feasibility: Participant Engagement
Description: Demonstrate that the delivery of the intervention(s) and the control intervention(s) under study can be delivered consistently, as defined by: 85% or more of randomized participants engage in 1 or more sessions; 75% or more of randomized participants engage in at least 6 of 9 sessions
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Partners4Pain Program | Key to Wellbeing Program
Number analyzed (Participants) | 26 | 25
Participants
  Engage in 1 or more sessions | 24 | 25
  Engage in 6 or more sessions | 24 | 24

5. Primary Outcome: Intervention Fidelity: Facilitator Delivery of Required Activities
Description: Demonstrate the fidelity of the intervention(s) used in the study by: Program facilitators deliver 90% of session activities during at least 90% of sessions
Time Frame: 9 weeks
Measure: Count of Units; unit: Sessions
Units Other Than Participants: Sessions
Arm/Group | Partners4Pain Program | Key to Wellbeing Program
Number analyzed (Participants) | 26 | 25
Number analyzed (Sessions) | 9 | 9
Sessions | 9 | 9

6. Primary Outcome: Data Collection Feasibility: Completion of Self-reported Outcomes
Description: Demonstrate the ability to collect study data by: 80% or more of randomized participants complete follow up at 2 months (end of the study)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Partners4Pain Program | Key to Wellbeing Program
Number analyzed (Participants) | 26 | 25
Participants | 24 | 25

7. Primary Outcome: Safety and Tolerability of the Interventions: Severe or Serious Related Adverse Events
Description: Demonstrate the safety and tolerability of the intervention(s) used in the study by: 5% or less of randomized participants experience a severe or serious adverse event related to the interventions
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Partners4Pain Program | Key to Wellbeing Program
Number analyzed (Participants) | 26 | 25
Participants | 0 | 1

8. Primary Outcome: Safety and Tolerability of the Interventions: Satisfaction With Program
Description: Demonstrate the safety and tolerability of the intervention(s) used in the study by: 75% or more of randomized participants are satisfied with assigned program
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Partners4Pain Program | Key to Wellbeing Program
Number analyzed (Participants) | 26 | 25
Participants | 21 | 21

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Partners4Pain Program | Key to Wellbeing Program
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/25
Other Adverse Events (participants affected / at risk) | 8/26 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partners4Pain Program (N=26) | Key to Wellbeing Program (N=25)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partners4Pain Program (N=26) | Key to Wellbeing Program (N=25)
Worsening back or neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Increased muscle soreness (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Feeling more upset than usual when reminded of the past (Psychiatric disorders) | 2 (2) | 2 (2)
Increased feelings of sadness (Psychiatric disorders) | 3 (3) | 2 (2)
Increased feelings of anxiousness (Psychiatric disorders) | 2 (2) | 4 (4)
Feeling more tired or fatigued than usual (General disorders) | 3 (3) | 8 (8)
Feeling more isolated or lonely (Social circumstances) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT05786508/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05786508/ICF_000.pdf